CLINICAL TRIAL: NCT03627195
Title: A Randomized, Double Blind, Placebo Controlled, Single Ascending Dose Study With Lurasidone Injectable Suspension to Evaluate Safety, Tolerability and Pharmacokinetics in Subjects With Schizophrenia
Brief Title: A Study to Determine the Maximum Tolerated Dose of an Investigational Drug in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1052024
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DSP-1349M (Experimental): Lurasidone injection suspension (30 mg, 75 mg, 150 mg, 300 mg, and 450 mg)
  Interventions: Drug: DSP-1349M
- Placbo (Placebo Comparator): placebo injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DSP-1349M — DSP-1349M injectable
  Other Names: lurasidone
  Arms: DSP-1349M
Drug: placebo — placebo injection
  Arms: Placbo

SUMMARY:
A study to determine the maximum tolerated dose of an investigational drug in subjects with schizophrenia

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, inpatient, single ascending dose (SAD) study designed to evaluate the safety, tolerability, and PK of lurasidone injectable suspension in subjects with schizophrenia. This study will determine the minimum intolerable dose (MID), the maximum tolerated dose (MTD) of lurasidone injectable suspension, and characterize the PK profiles of lurasidone and its metabolites in serum (ID-14283, ID-14326, ID-11614, ID-20219, and ID-20220) and urine (ID-14283, ID-14326, and ID-11614) in this subject population. The potential effects of gender on the PK of lurasidone injectable suspension and its metabolites will also be evaluated when applicable.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject has capacity; is willing and able to provide written consent for use and disclosure of protected health information per requirements of 45CFR164.508 (Health Insurance Portability and Accountability Act; HIPAA) prior to initiating any study procedure after being informed of the nature of the study, in the opinion of the study staff and PI.

  2. Subject is male or female 18 to 65 years of age, inclusive. 3. Subject has a diagnosis of schizophrenia as per DSM-IV-TR criteria, which in the opinion of the Investigator has been clinically stable for the past 6 months.

  4. Subject has a Body Mass Index (BMI) greater than or equal to 19.5 and less than or equal to 38 kg/m2.

  5. Subject does not have clinically relevant abnormal laboratory values per Investigator discretion.

  6. Subject does not have clinically relevant findings from vital signs measurements per Investigator discretion.

  7. Female subject is eligible to enter and participate in the study if she is of:

  a. Non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal);
* Postmenopausal females defined as being amenorrheic for greater than 2 years (or confirmed by FSH level) with an appropriate clinical profile.
* Women who have not been confirmed as postmenopausal should be advised to use contraception as outlined below.
* Women who have had a hysterectomy, bilateral oophorectomy or bilateral salpingectomy (as determined by subject's medical history).

  b. Child-bearing potential (all females ≤ 65 years of age), has a negative pregnancy test at screening and agrees to satisfy one of the following requirements:
* Complete abstinence from intercourse (as part of an abstinent lifestyle) a minimum of 2 months prior to administration of the first dose of study drug, throughout the Treatment Period, and for a minimum of 3 months after completion or premature discontinuation from the study drug; or,
* Established use of highly effective methods of contraception from 1 month prior to administration of the first dose of study drug, during the Treatment Period, and 60 days after completion or premature discontinuation from the study drug.

  * Because of the unacceptable failure rate of barrier (chemical and/or physical) methods, the barrier method of contraception must only be used in combination with a highly effective method. Post-coital methods of contraception are not permitted.

    8. Male subjects with partners of child bearing potential must be practicing abstinence, part of an abstinent life style or using protocol-specified methods of birth control throughout the study and for 30 days after completion or premature discontinuation from the study drug.

    9. Subject is able and willing to remain off of prior antipsychotic medication until the protocol-specified restabilization period.

    10. Subject has a stable living arrangement for at least 3 months prior to Day -12 and agrees to return to a similar living arrangement after discharge. Such subjects remain eligible to participate in this protocol with approval from the PI. Chronically homeless subjects should not be enrolled. The Medical Monitor should be consulted for individual cases as

Exclusion Criteria:

1. Subject had an acute exacerbation of psychiatric symptoms requiring change in antipsychotic medication (with reference to drug or dose) within 3 months (90 days) before screening.
2. Subject has known or suspected carcinoma.
3. Subject has known presence or history of renal or hepatic insufficiency.
4. Subject has significant disease(s) or clinically significant finding(s) on physical examination determined by the Investigator to pose a health concern to the subject while on study.
5. Subject has a history or presence of clinically significant abnormal ECG (based on ECG central overread report) that may jeopardize the subject's safety to participate in this study, or a screening 12-lead ECG demonstrating any one of the following: heart rate (HR) > 100 bpm, QRS > 120 msec, QTcF > 450 msec, or PR > 220 msec.
6. Subject has known history of a severe reaction to a previous antipsychotic (in the Investigator's opinion), including up to 80 mg/day of oral lurasidone.
7. Subject has a history of drug-dependence as per DSM-IV-TR criteria during the six month period immediately prior to study entry.
8. Subject has known or suspected excessive alcohol consumption, (exceeding more than 4 drinks on any single day or more than 14 drinks per week; 1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of the screening visit or a positive urine alcohol test at screening.
9. Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS at screening (in the past 1 month [30 days]) or at any point prior to randomization or history of suicidal behavior within the last two years.
10. Subject has significant orthostatic hypotension at screening (ie, a drop in systolic blood pressure of 30 mmHg or more and/or drop in diastolic blood pressure of 20 mmHg or more on standing).
11. Subject has presence or history (within the last year) of a medical or surgical condition that might interfere with the absorption, metabolism, or excretion of administered Lurasidone injectable suspension.
12. Subject has a history of epilepsy or risk of having seizures.
13. Subject has a positive urine alcohol at screening or on Day -12.
14. Subject has positive test results within 28 days prior to the start of the study for:

    1. Human immunodeficiency virus (HIV).
    2. Hepatitis B surface antigen and Hepatitis C antibody.
    3. Urine drug test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, methadone, or other drugs of abuse). However, a positive test for benzodiazepines may not result in exclusion of subjects if the Investigator determines that the use of a prescription benzodiazepine is appropriate.
    4. Serum β-human chorionic gonadotropin (HCG) consistent with pregnancy (females only).
15. Subject has used of any inhibitor or inducer of CYP3A4 taken within 28 days prior to drug administration and until discharge.
16. Subject has have used of concomitant medications that prolong the QT/QTc interval within 28 days prior to Day -12 through follow-up.
17. Subject has received depot neuroleptics unless the last injection was at least one treatment cycle before Day -12.
18. Subject has poor peripheral venous access or does not tolerate venipuncture that would cause difficulty for collecting blood samples.
19. Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 30 days prior to screening, or intends to donate plasma or blood or undergo elective surgery during study participation or within 30 days after the last study visit.
20. Subject has a prolactin concentration greater than or equal to 200 ng/mL at screening.
21. Subject is unwilling to abstain from vigorous exercise from Day -12 until study discharge.
22. Subjects has a significant risk of violent behavior or a significant risk of suicidal behavior based on history or in the PI's judgment OR is considered by the Investigator to be at imminent risk of suicide or injury to self, others, or property.
23. Subject has a history of allergic reaction (clinically relevant history of drug hypersensitivity) or has a known or suspected sensitivity to any substance that is contained in the study drug or to Polysorbate 80, sodium chloride, or sodium phosphate.
24. Subject requires treatment with a drug that consistently prolongs the QTc interval.
25. Subject is currently participating, or has participated in a study with an investigational or marketed compound or device within 30 days prior to signing the informed consent, or Protocol D1052024, Version 2.00 Lurasidone Injectable Suspension Confidential and Proprietary 36 13 June 2018 has participated in 3 or more studies within 18 months prior to signing the informed consent.
26. Subject is a staff member or the relative of a staff member.
27. Subject, in the Investigator's opinion, is unsuitable in any other way to participate in the study.
28. Subject is unable or unwilling to comply with study instructions, procedures or restrictions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. David Walling, Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 30 mg: Lurasidone injection suspension 30 mg
- Lurasidone 75 mg: Lurasidone injection suspension 75 mg
- Lurasidone 150 mg: Lurasidone injection suspension 150 mg
- Lurasidone 300 mg: Lurasidone injection suspension 300 mg
- Lurasidone 450 mg: Lurasidone injection suspension 450 mg
Period: Overall Study
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 5 | 6 | 6 | 6 | 6 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — OTHER (LACK OF EFFICACY) | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (13.29) | 45 (10.22) | 52 (4.47) | 46.2 (9.72) | 52.8 (11.81) | 45.7 (10.25) | 47.4 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 1 | 5 | 15
  Male | 3 | 4 | 4 | 4 | 5 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 0 | 2 | 6
  Not Hispanic or Latino | 5 | 5 | 6 | 4 | 6 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 5 | 4 | 5 | 4 | 4 | 7 | 29
  White | 1 | 2 | 1 | 1 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 170 (8.83) | 173.2 (8.61) | 174.3 (10.39) | 166.3 (7.92) | 174.2 (7.25) | 168.5 (7.07) | 170.8 (8.29)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 88.3 (13.53) | 80.3 (10.86) | 84.8 (21.84) | 82 (16.55) | 86.8 (15.2) | 86.7 (15.07) | 85 (14.99)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.88 (6.444) | 27.1 (5.522) | 27.68 (5.975) | 29.83 (6.493) | 28.77 (5.125) | 30.37 (3.919) | 29.23 (5.295)
Baseline Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) Total Score is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210 Higher values of PANSS total score represents greater severity of illness.
  units on a scale | 60.2 (7.76) | 62 (8.25) | 59.3 (7.94) | 53.7 (7.55) | 58.3 (6.8) | 64.3 (7.56) | 60.1 (7.93)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events (AEs ) Leading to Study Discontinuation
Description: Number of subjects with any Adverse Events (AEs), serious adverse events (SAEs), and Adverse Events (AEs ) leading to study discontinuation
Time Frame: Day 61
Measure: Number; unit: count of participants
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
count of participants
  Incidence of AEs | 4 | 4 | 2 | 4 | 5 | 5
  Incidence of SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Incidence of AEs leading to study discontinuation | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Serum Concentration [Cmax] for Lurasidone After Lurasidone Injectable Suspension Administration
Description: The maximum Serum Concentration [Cmax] for lurasidone after lurasidone injectable suspension administration
Time Frame: Day 61
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 10
ng/mL | 1.08 (65.6) | 3.90 (51.6) | 5.08 (46.5) | 8.85 (62.8) | 9.50 (48.3) | 0 (0)

3. Primary Outcome: Area Under the Curve From Time 0 to Time of Last Quantifiable Concentration [AUC0-last] for Lurasidone After Lurasidone Injectable Suspension Administration
Description: The area Under the Curve from time 0 to time of last quantifiable concentration [AUC0-last] for lurasidone after lurasidone injectable suspension administration
Time Frame: Day 61
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 10
ng*h/mL | 628 (54.7) | 2000 (6.6) | 3540 (26.0) | 4910 (47.9) | 7490 (32.6) | 0 (0)

ADVERSE EVENTS:
Time Frame: 61 days
Arm/Group | Lurasidone 30 mg | Lurasidone 75 mg | Lurasidone 150 mg | Lurasidone 300 mg | Lurasidone 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 4/6 | 5/6 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 30 mg (N=6) | Lurasidone 75 mg (N=6) | Lurasidone 150 mg (N=6) | Lurasidone 300 mg (N=6) | Lurasidone 450 mg (N=6) | Placebo (N=10)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postural tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT03627195/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03627195/SAP_001.pdf